CLINICAL TRIAL: NCT07328425
Title: Phase II Study of Lurbinectedin and Irinotecan in Adult and Young Adult Patients With Advanced Desmoplastic Small Round Cell Tumor (DSRCT)
Brief Title: Clinical Study in Patients With DSRCT
Acronym: ISG-TULIPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISG-TULIPS; 2024-519261-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Desmoplastic Small Round Cell Tumor
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor | interventions — PM 01183; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lurbinectedine and Irinotecan (Experimental): lurbinectedin in combination with intravenous irinotecan administered until progression or unacceptable toxicity, in a population of =/>15 years old patients with histologically and molecularly confirmed (EWSR1-WT1 translocation positive), advanced (locally advanced or metastatic) DSRCT, from 2nd to 4th line, following progression to anthracycline-based chemotherapy.
  Interventions: Drug: Lurbinectedin; Drug: Irinotecan

INTERVENTIONS:
Drug: Lurbinectedin — Lurbinectedin and Irinotecan
Drug: Irinotecan — Lurbinectedin and Irinotecan

SUMMARY:
Patients participating in this study have DSRCT that has spread locally or to other parts of the body and can no longer be surgically removed without causing significant harm.

Treatment will continue until the tumor progresses further, severe side effects occur, or either patient or investigator decision.

In addition, patients may participate in an optional biological study. The study will analyze the tumor's genes and the molecules related to them. By studying genes and their products, the investigators can better understand the behavior of the tumor and how the body responds to therapies.

DETAILED DESCRIPTION:
This is an Italian and Spanish multicentric, prospective, phase II single-arm, open-label, investigator-initiated clinical study that will be conducted within the Italian Sarcoma Group (ISG) and the Spanish Sarcoma Groups (GEIS), aiming at exploring the activity of lurbinectedinin combination with irinotecan, until progression or unacceptable toxicity, in a population of =/>15 years old patients with histologically and molecularly confirmed (EWSR1-WT1 translocation positive), advanced (locally advanced or metastatic) DSRCT, from 2nd to 4th line, following progression to anthracycline-based chemotherapy.

The primary end-point of the study will be the overall response rate (ORR) by RECIST v1.1 in the study population. Secondary end-points will be PFS, DoR, OS, safety and changes in QoL.

Patients will be evaluated for the primary end-point if have completed at least one cycle of lurbinectedin and irinotecan and have at least one post-baseline radiologic disease assessment. Patients with documented early progression disease (PD) or who die due to PD before the first scheduled tumor assessment will also be included in the analysis.

Patients will be followed for follow up visits every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histological centrally confirmed diagnosis of DSRCT with the documented presence of EWSR1-WT1 translocation.
2. Age ≥ 15 years.
3. Locally advanced (i.e. radical surgical resection of local disease unfeasible or surgery declined by the patient or surgery deemed to become less demolitive and / or easier after cytoreduction) and/or metastatic disease.
4. Measurable disease by RECIST v1.1.
5. Clinical or objective disease progression after the last administration of the last standard therapy, or have stopped standard therapy due to intolerability within 6 months from enrollment.
6. At least one prior chemotherapy based on anthracycline (considering chemotherapy administered for primary tumour) and no more than 3 prior chemotherapy lines.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2.
8. Adequate bone marrow, renal, hepatic, and metabolic function (assessed ≤ 7 days before inclusion in the trial), defined as the following:

   1. platelet count ≥ 100 × 109/L, hemoglobin ≥ 9.0 g/dL, white blood cells ≥ 3.0 × 109/L and absolute neutrophil count (ANC) ≥ 2.0 × 109/L,
   2. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × the upper limit of normal (ULN), even in the presence of liver metastases,
   3. total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤ ULN,
   4. International Normalized Ratio (INR) < 1.5 (except if patient is on oral anticoagulation therapy),
   5. calculated creatinine clearance (CrCL) ≥ 30 mL/minute (using Cockcroft-Gault formula),
   6. creatine phosphokinase (CPK) ≤ 2.5 × ULN,
   7. albumin ≥ 3.0 g/dL.
9. Cardiac ejection fraction ≥50% as measured by echocardiogram.
10. Recovery to grade ≤ 1 or to baseline from any adverse event (AE) derived from previous treatment (excluding alopecia and/or cutaneous toxicity and/or fatigue grade ≤ 2).
11. No history of arterial and/or venous thromboembolic event within the previous 12 months.
12. Females of childbearing potential must have a negative pregnancy test (preferable by serum or, if serum test unavailable, urine beta-HCG) within 7 days before treatment start.
13. Post-menopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential.
14. Male and female patients of reproductive potential must agree to employ a highly effective method of birth control (Acceptable methods of contraception are described in Appendix 5) throughout the study and thereafter, at the end of study treatment, and for at least 7 months from the patient's last lurbinectedin administration in female patients of childbearing potential and for at least 4 months in men in fertile age after the last lurbinectedin administration.
15. The patient or legal representative must be able to read and understand the informed consent form (ICF) and must have been willing to give written informed consent and any locally required authorisation before any study-specific procedures, including screening evaluations, sampling, and analyses.

Exclusion Criteria:

1. Prior treatment with lurbinectedin or trabectedin, Ecubectedin (PM 14) or PM54.
2. Known hypersensitivity to irinotecan or lurbinectedin or any of their components of the drugs products (excipients).
3. Other primary malignancy with <5 years clinically assessed disease free interval, except basal cell skin cancer, cervical carcinoma in situ or other neoplasm judged to entail a low risk of relapse.
4. History or presence of unstable angina, myocardial infarction, or clinically significant valvular heart disease within 12 months of the study.
5. Grade III/IV cardiac problems as defined by the New York Heart Association Criteria (i.e. congestive heart failure, myocardial infarction within 12 months of study).
6. Symptomatic arrhythmia or any uncontrolled arrhythmia requiring ongoing treatment within 12 months of study.
7. Myopathy or any clinical situation that causes significant and persistent elevation of CPK (> 2.5 × ULN in two different determinations performed one week apart).
8. Severe and/or uncontrolled medical disease (i.e. uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
9. Known active brain metastasis.
10. Known chronic liver disease (i.e. chronic active hepatitis and cirrhosis).
11. Diagnosis of human deficiency virus (HIV), hepatitis C virus (HCV) infection or active hepatitis B (to be excluded during the screening period).
12. Any past or present chronic inflammatory colon and/or liver disease, past intestinal obstruction, pseudo or sub-occlusion or paralysis.
13. Evident symptomatic pulmonary fibrosis or interstitial pneumonitis, pleural or cardiac effusion rapidly increasing and/or necessitating prompt local treatment within seven days.
14. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
15. Known active COVID-19 disease (this includes positive test for SARS-CoV-2 in nasopharyngeal/oropharyngeal swabs or nasal swabs by PCR).
16. Prior bone marrow and/or stem cell transplantation, and allogenic transplant.
17. Last dose of systemic cytotoxic therapy or investigational therapy within 21 days from enrollment.
18. Prior treatment with any form of radiation therapy within 14 days from enrollment.
19. Major surgery within 3 weeks prior to study entry and minor surgery within 1 week prior to study entry.
20. Use of strong inducers of CYP3A activity within two weeks prior to the first infusion of lurbinectedin (Appendix 6).
21. Expected limitation of the patient's ability to comply with the treatment or follow-up protocol.
22. Subjects who have current active hepatic or biliary disease (with exception of patients with asymptomatic gallstones, liver metastasis or stable chronic liver disease per Investigator assessment).
23. Subjects who have known Gilbert's syndrome.
24. Patient has received a live or liver attenuated vaccines within 30 days before the first dose of study intervention. Killed vaccines are allowed.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall tumour Response Rate (ORR), according to RECIST v 1.1 | Week 6, week 12, week 18, week 30, week 42, week 54, week 66, week 78, week 90, week 102 and until progression
  Overall tumour Response Rate (ORR), according to RECIST v 1.1

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of study therapy start until the date of death from any cause, assessed up to 60 months
  Overall Survival (OS)
Progression Free Survival (PFS) | From date of study therapy start until first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression Free Survival (PFS)
Duration of Response (DoR) | From date of study therapy start until first documented assessment without progression or date of death from any cause, whichever came first, assessed up to 60 months
  Duration of Response (DoR)
Adverse events and Serious adverse event (according to CTC-AE v.5) | After initiation of study treatments(s), all adverse events will be reported until 30 days after the final dose of study treatment or until initiation of new systemic anti-cancer therapy, whichever occurs first.
  Adverse events and Serious adverse event (according to CTC-AE v.5)
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Screening, cycle1 day1 (each cycle is 21 days), cycle2 day1, End Of Treatment visit (performed 30 days after the last study drug administration), at follow-up visits performed at months 6, 12, 18 and 24 after the last study drug administration
  The EORTC QLQ-C30 is a validated 30-item questionnaire assessing health-related quality of life in cancer patients. Scores are linearly transformed to a 0 to 100 scale.
  For the Global Health Status/Quality of Life and functional scales (physical, role, emotional, cognitive, and social functioning), higher scores indicate better quality of life or functioning.
  For the symptom scales and single-item symptom measures, higher scores indicate greater symptom severity (worse outcome).
Brief Inventory Pain questionnaire | Screening, cycle1 day1 (each cycle is 21 days), cycle2 day1, End Of Treatment visit (performed 30 days after the last study drug administration), at follow-up visits performed at months 6, 12, 18 and 24 after the last study drug administration
  Brief Inventory Pain questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Syecchiotti, MD, Principal Investigator — Findazione IRCCS Istituto Nazionale Tumori Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jayakrishnan T, Moll R, Sandhu A, Sanguino A, Kaur G, Mao S. Desmoplastic Small Round-cell Tumor: Retrospective Review of Institutional Data and Literature Review. Anticancer Res. 2021 Aug;41(8):3859-3866. doi: 10.21873/anticanres.15179. PMID 34281846
- [Background] Hayes-Jordan AA, Coakley BA, Green HL, Xiao L, Fournier KF, Herzog CE, Ludwig JA, McAleer MF, Anderson PM, Huh WW. Desmoplastic Small Round Cell Tumor Treated with Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy: Results of a Phase 2 Trial. Ann Surg Oncol. 2018 Apr;25(4):872-877. doi: 10.1245/s10434-018-6333-9. Epub 2018 Jan 30. PMID 29383611
- [Background] Rosoff PM, Bayliff S. Successful clinical response to irinotecan in desmoplastic round blue cell tumor. Med Pediatr Oncol. 1999 Nov;33(5):500-3. doi: 10.1002/(sici)1096-911x(199911)33:53.0.co;2-x. No abstract available. PMID 10531577
- [Background] Honore C, Amroun K, Vilcot L, Mir O, Domont J, Terrier P, Le Cesne A, Le Pechoux C, Bonvalot S. Abdominal desmoplastic small round cell tumor: multimodal treatment combining chemotherapy, surgery, and radiotherapy is the best option. Ann Surg Oncol. 2015 Apr;22(4):1073-9. doi: 10.1245/s10434-014-4123-6. Epub 2014 Oct 10. PMID 25300608
- [Background] Stacchiotti S, Frezza AM, Blay JY, Baldini EH, Bonvalot S, Bovee JVMG, Callegaro D, Casali PG, Chiang RC, Demetri GD, Demicco EG, Desai J, Eriksson M, Gelderblom H, George S, Gounder MM, Gronchi A, Gupta A, Haas RL, Hayes-Jardon A, Hohenberger P, Jones KB, Jones RL, Kasper B, Kawai A, Kirsch DG, Kleinerman ES, Le Cesne A, Lim J, Chirlaque Lopez MD, Maestro R, Marcos-Gragera R, Martin Broto J, Matsuda T, Mir O, Patel SR, Raut CP, Razak ARA, Reed DR, Rutkowski P, Sanfilippo RG, Sbaraglia M, Schaefer IM, Strauss DC, Sundby Hall K, Tap WD, Thomas DM, van der Graaf WTA, van Houdt WJ, Visser O, von Mehren M, Wagner AJ, Wilky BA, Won YJ, Fletcher CDM, Dei Tos AP, Trama A. Ultra-rare sarcomas: A consensus paper from the Connective Tissue Oncology Society community of experts on the incidence threshold and the list of entities. Cancer. 2021 Aug 15;127(16):2934-2942. doi: 10.1002/cncr.33618. Epub 2021 Apr 28. PMID 33910263
- [Background] Saab R, Khoury JD, Krasin M, Davidoff AM, Navid F. Desmoplastic small round cell tumor in childhood: the St. Jude Children's Research Hospital experience. Pediatr Blood Cancer. 2007 Sep;49(3):274-9. doi: 10.1002/pbc.20893. PMID 16685737
- [Background] Liu KX, Collins NB, Greenzang KA, Furutani E, Campbell K, Groves A, Mullen EA, Shusterman S, Spidle J, Marcus KJ, Weil BR, Weldon CB, Frazier AL, Janeway KA, O'Neill AF, Mack JW, DuBois SG, Shulman DS. The use of interval-compressed chemotherapy with the addition of vincristine, irinotecan, and temozolomide for pediatric patients with newly diagnosed desmoplastic small round cell tumor. Pediatr Blood Cancer. 2020 Oct;67(10):e28559. doi: 10.1002/pbc.28559. Epub 2020 Jul 19. PMID 32686305
- [Background] Verret B, Honore C, Dumont S, Terrier P, Adam J, Cavalcanti A, Sourrouille I, Klausner G, Ahlenc-Gelas M, Kiavue N, Domitrescu G, El Amarti L, Mir O, Le Cesne A. Trabectedin in advanced desmoplastic round cell tumors: a retrospective single-center series. Anticancer Drugs. 2017 Jan;28(1):116-119. doi: 10.1097/CAD.0000000000000435. PMID 27782906
- [Background] Giani C, Radaelli S, Miceli R, Gandola L, Sangalli C, Frezza AM, Provenzano S, Pasquali S, Bertulli R, Fiore M, Callegaro D, Casanova M, Chiaravalli S, Collini P, Dagrada GP, Morosi C, Zaffaroni N, Casali PG, Ferrari A, Gronchi A, Stacchiotti S. Long-term survivors with desmoplastic small round cell tumor (DSRCT): Results from a retrospective single-institution case series analysis. Cancer Med. 2023 May;12(9):10694-10703. doi: 10.1002/cam4.5829. Epub 2023 Mar 23. PMID 36951537
- [Background] Brunetti AE, Delcuratolo S, Lorusso V, Palermo L, Di Giorgio A, Pisconti S, Silvestris N. Third-line trabectedin for a metastatic desmoplastic small round cell tumour treated with multimodal therapy. Anticancer Res. 2014 Jul;34(7):3683-8. PMID 24982387
- [Background] Leal JF, Martinez-Diez M, Garcia-Hernandez V, Moneo V, Domingo A, Bueren-Calabuig JA, Negri A, Gago F, Guillen-Navarro MJ, Aviles P, Cuevas C, Garcia-Fernandez LF, Galmarini CM. PM01183, a new DNA minor groove covalent binder with potent in vitro and in vivo anti-tumour activity. Br J Pharmacol. 2010 Nov;161(5):1099-110. doi: 10.1111/j.1476-5381.2010.00945.x. PMID 20977459
- [Background] Lettieri CK, Garcia-Filion P, Hingorani P. Incidence and outcomes of desmoplastic small round cell tumor: results from the surveillance, epidemiology, and end results database. J Cancer Epidemiol. 2014;2014:680126. doi: 10.1155/2014/680126. Epub 2014 Nov 5. PMID 25431592
- [Background] Zuco V, Pasquali S, Tortoreto M, Percio S, Doldi V, Barisella M, Collini P, Dagrada GP, Brich S, Gasparini P, Fiore M, Casanova M, Frezza AM, Gronchi A, Stacchiotti S, Ferrari A, Zaffaroni N. Effectiveness of irinotecan plus trabectedin on a desmoplastic small round cell tumor patient-derived xenograft. Dis Model Mech. 2023 Jun 1;16(6):dmm049649. doi: 10.1242/dmm.049649. Epub 2023 Jun 14. PMID 37158111
- [Background] Scheer M, Vokuhl C, Blank B, Hallmen E, von Kalle T, Munter M, Wessalowski R, Hartwig M, Sparber-Sauer M, Schlegel PG, Kramm CM, Kontny U, Spriewald B, Kegel T, Bauer S, Kazanowska B, Niggli F, Ladenstein R, Ljungman G, Jahnukainen K, Fuchs J, Bielack SS, Klingebiel T, Koscielniak E; Cooperative Weichteilsarkom Studiengruppe [CWS]. Desmoplastic small round cell tumors: Multimodality treatment and new risk factors. Cancer Med. 2019 Feb;8(2):527-542. doi: 10.1002/cam4.1940. Epub 2019 Jan 16. PMID 30652419
- [Background] Stiles ZE, Dickson PV, Glazer ES, Murphy AJ, Davidoff AM, Behrman SW, Bishop MW, Martin MG, Deneve JL. Desmoplastic small round cell tumor: A nationwide study of a rare sarcoma. J Surg Oncol. 2018 Jun;117(8):1759-1767. doi: 10.1002/jso.25071. Epub 2018 Jun 7. PMID 29878371
- [Background] Italiano A, Kind M, Cioffi A, Maki RG, Bui B. Clinical activity of sunitinib in patients with advanced desmoplastic round cell tumor: a case series. Target Oncol. 2013 Sep;8(3):211-213. doi: 10.1007/s11523-012-0251-8. Epub 2013 Jan 6. PMID 23292310
- [Background] Van Glabbeke M, Verweij J, Judson I, Nielsen OS; EORTC Soft Tissue and Bone Sarcoma Group. Progression-free rate as the principal end-point for phase II trials in soft-tissue sarcomas. Eur J Cancer. 2002 Mar;38(4):543-9. doi: 10.1016/s0959-8049(01)00398-7. PMID 11872347
- [Background] Bisogno G, Ferrari A, Tagarelli A, Sorbara S, Chiaravalli S, Poli E, Scarzello G, De Corti F, Casanova M, Affinita MC. Integrating irinotecan in standard chemotherapy: A novel dose-density combination for high-risk pediatric sarcomas. Pediatr Blood Cancer. 2021 Jul;68(7):e28951. doi: 10.1002/pbc.28951. Epub 2021 Mar 10. PMID 33694265
- [Background] Frezza AM, Whelan JS, Dileo P. Trabectedin for desmoplastic small round cell tumours: a possible treatment option? Clin Sarcoma Res. 2014 Apr 25;4:3. doi: 10.1186/2045-3329-4-3. eCollection 2014. PMID 24829745
- [Background] Harlow ML, Chasse MH, Boguslawski EA, Sorensen KM, Gedminas JM, Kitchen-Goosen SM, Rothbart SB, Taslim C, Lessnick SL, Peck AS, Madaj ZB, Bowman MJ, Grohar PJ. Trabectedin Inhibits EWS-FLI1 and Evicts SWI/SNF from Chromatin in a Schedule-dependent Manner. Clin Cancer Res. 2019 Jun 1;25(11):3417-3429. doi: 10.1158/1078-0432.CCR-18-3511. Epub 2019 Feb 5. PMID 30723142
- [Background] Lima M, Bouzid H, Soares DG, Selle F, Morel C, Galmarini CM, Henriques JA, Larsen AK, Escargueil AE. Dual inhibition of ATR and ATM potentiates the activity of trabectedin and lurbinectedin by perturbing the DNA damage response and homologous recombination repair. Oncotarget. 2016 May 3;7(18):25885-901. doi: 10.18632/oncotarget.8292. PMID 27029031
- [Background] Harlow ML, Maloney N, Roland J, Guillen Navarro MJ, Easton MK, Kitchen-Goosen SM, Boguslawski EA, Madaj ZB, Johnson BK, Bowman MJ, D'Incalci M, Winn ME, Turner L, Hostetter G, Galmarini CM, Aviles PM, Grohar PJ. Lurbinectedin Inactivates the Ewing Sarcoma Oncoprotein EWS-FLI1 by Redistributing It within the Nucleus. Cancer Res. 2016 Nov 15;76(22):6657-6668. doi: 10.1158/0008-5472.CAN-16-0568. Epub 2016 Oct 3. PMID 27697767
- [Background] Bailey K, Roth M, Weiser D, Gill J. High-Dose Chemotherapy with Stem Cell Rescue in Desmoplastic Small Round Cell Tumor: A Single-Institution Experience and Review of the Literature. Sarcoma. 2018 May 6;2018:1948093. doi: 10.1155/2018/1948093. eCollection 2018. PMID 29853779
- [Background] Lopez-Gonzalez A, Cantos B, Tejerina E, Provencio M. Activity of trabectidin in desmoplastic small round cell tumor. Med Oncol. 2011 Dec;28 Suppl 1:S644-6. doi: 10.1007/s12032-010-9687-9. Epub 2010 Oct 7. PMID 20924717
- [Background] Mello CA, Campos FAB, Santos TG, Silva MLG, Torrezan GT, Costa FD, Formiga MN, Nicolau U, Nascimento AG, Silva C, Curado MP, Nakagawa SA, Lopes A, Aguiar S Jr. Desmoplastic Small Round Cell Tumor: A Review of Main Molecular Abnormalities and Emerging Therapy. Cancers (Basel). 2021 Jan 28;13(3):498. doi: 10.3390/cancers13030498. PMID 33525546
- [Background] Ferreira EN, Barros BD, de Souza JE, Almeida RV, Torrezan GT, Garcia S, Krepischi AC, Mello CA, Cunha IW, Pinto CA, Soares FA, Dias-Neto E, Lopes A, de Souza SJ, Carraro DM. A genomic case study of desmoplastic small round cell tumor: comprehensive analysis reveals insights into potential therapeutic targets and development of a monitoring tool for a rare and aggressive disease. Hum Genomics. 2016 Nov 18;10(1):36. doi: 10.1186/s40246-016-0092-0. PMID 27863505
- [Background] Devecchi A, De Cecco L, Dugo M, Penso D, Dagrada G, Brich S, Stacchiotti S, Sensi M, Canevari S, Pilotti S. The genomics of desmoplastic small round cell tumor reveals the deregulation of genes related to DNA damage response, epithelial-mesenchymal transition, and immune response. Cancer Commun (Lond). 2018 Nov 28;38(1):70. doi: 10.1186/s40880-018-0339-3. PMID 30486883
- [Background] Frezza AM, Benson C, Judson IR, Litiere S, Marreaud S, Sleijfer S, Blay JY, Dewji R, Fisher C, van der Graaf W, Hayward L. Pazopanib in advanced desmoplastic small round cell tumours: a multi-institutional experience. Clin Sarcoma Res. 2014 Jul 29;4:7. doi: 10.1186/2045-3329-4-7. eCollection 2014. PMID 25089183
- [Background] Santiago L, Daniels G, Wang D, Deng FM, Lee P. Wnt signaling pathway protein LEF1 in cancer, as a biomarker for prognosis and a target for treatment. Am J Cancer Res. 2017 Jun 1;7(6):1389-1406. eCollection 2017. PMID 28670499
- [Background] Gedminas JM, Kaufman R, Boguslawski EA, Gross AC, Adams M, Beddows I, Kitchen-Goosen SM, Roberts RD, Grohar PJ. Lurbinectedin Inhibits the EWS-WT1 Transcription Factor in Desmoplastic Small Round Cell Tumor. Mol Cancer Ther. 2022 Aug 2;21(8):1296-1305. doi: 10.1158/1535-7163.MCT-21-1003. PMID 35657345
- [Background] Bisogno G, Ferrari A, Rosolen A, Alaggio R, Scarzello G, Garaventa A, Arcamone G, Carli M. Sequential intensified chemotherapy with stem cell rescue for children and adolescents with desmoplastic small round-cell tumor. Bone Marrow Transplant. 2010 May;45(5):907-11. doi: 10.1038/bmt.2009.248. Epub 2009 Oct 5. PMID 19802018
- [Background] Di Maio M, Basch E, Bryce J, Perrone F. Patient-reported outcomes in the evaluation of toxicity of anticancer treatments. Nat Rev Clin Oncol. 2016 May;13(5):319-25. doi: 10.1038/nrclinonc.2015.222. Epub 2016 Jan 20. PMID 26787278
- [Background] Uboldi S, Craparotta I, Colella G, Ronchetti E, Beltrame L, Vicario S, Marchini S, Panini N, Dagrada G, Bozzi F, Pilotti S, Galmarini CM, D'Incalci M, Gatta R. Mechanism of action of trabectedin in desmoplastic small round cell tumor cells. BMC Cancer. 2017 Feb 6;17(1):107. doi: 10.1186/s12885-017-3091-1. PMID 28166781
- [Background] Ferrari A, Bergamaschi L, Chiaravalli S, Pecori E, Diletto B, Alessandro O, Giandini T, Livellara V, Sironi G, Casanova M. Multiagent chemotherapy including IrIVA regimen and maintenance therapy in the treatment of desmoplastic small round cell tumor. Tumori. 2022 Feb;108(1):93-97. doi: 10.1177/0300891621995250. Epub 2021 Feb 17. PMID 33594944
- [Background] Hayes-Jordan A, Green HL, Lin H, Owusu-Agyemang P, Fitzgerald N, Arunkumar R, Mejia R, Okhuysen-Cawley R, Mauricio R, Fournier K, Ludwig J, Anderson P. Complete cytoreduction and HIPEC improves survival in desmoplastic small round cell tumor. Ann Surg Oncol. 2014 Jan;21(1):220-4. doi: 10.1245/s10434-013-3269-y. Epub 2013 Sep 18. PMID 24046124
- [Background] Wei G, Shu X, Zhou Y, Liu X, Chen X, Qiu M. Intra-Abdominal Desmoplastic Small Round Cell Tumor: Current Treatment Options and Perspectives. Front Oncol. 2021 Sep 15;11:705760. doi: 10.3389/fonc.2021.705760. eCollection 2021. PMID 34604040
- [Background] Lal DR, Su WT, Wolden SL, Loh KC, Modak S, La Quaglia MP. Results of multimodal treatment for desmoplastic small round cell tumors. J Pediatr Surg. 2005 Jan;40(1):251-5. doi: 10.1016/j.jpedsurg.2004.09.046. PMID 15868593
- [Background] Romano M, Frapolli R, Zangarini M, Bello E, Porcu L, Galmarini CM, Garcia-Fernandez LF, Cuevas C, Allavena P, Erba E, D'Incalci M. Comparison of in vitro and in vivo biological effects of trabectedin, lurbinectedin (PM01183) and Zalypsis(R) (PM00104). Int J Cancer. 2013 Nov;133(9):2024-33. doi: 10.1002/ijc.28213. Epub 2013 May 25. PMID 23588839
- [Background] Ferrari A, Chiaravalli S, Bergamaschi L, Nigro O, Livellara V, Sironi G, Gasparini P, Pasquali S, Zaffaroni N, Stacchiotti S, Morosi C, Massimino M, Casanova M. Trabectedin-irinotecan, a potentially promising combination in relapsed desmoplastic small round cell tumor: report of two cases. J Chemother. 2023 Apr;35(2):163-167. doi: 10.1080/1120009X.2022.2067706. Epub 2022 Apr 26. PMID 35470779
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Hendricks A, Boerner K, Germer CT, Wiegering A. Desmoplastic Small Round Cell Tumors: A review with focus on clinical management and therapeutic options. Cancer Treat Rev. 2021 Feb;93:102140. doi: 10.1016/j.ctrv.2020.102140. Epub 2020 Dec 24. PMID 33388539